CLINICAL TRIAL: NCT00132431
Title: Sensipar Treatment Algorithm to Reach K/DOQI Targets in Chronic Kidney Disease Subjects With Secondary Hyperparathyroidism
Brief Title: START: Sensipar Treatment Algorithm to Reach K/DOQI Targets in Chronic Kidney Disease Subjects With Secondary Hyperparathyroidism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20040123
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Kidney Disease; Secondary Hyperparathyroidism; Chronic Kidney Disease
Keywords: calcimimetic; cinacalcet; hemodialysis; secondary hyperparathyroidism; chronic kidney disease
MeSH Terms: conditions — Kidney Diseases; Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic | interventions — Cinacalcet

INTERVENTIONS:
Drug: Sensipar

SUMMARY:
The purpose of this research is to study the effects and safety of Sensipar approved by the Food and Drug Administration (FDA) in patients with kidney failure who are being treated with dialysis and have uncontrolled secondary hyperparathyroidism (HPT).

DETAILED DESCRIPTION:
The purposes of this study are: - To assess the effectiveness of a treatment algorithm that includes Sensipar on bio-intact parathyroid hormone (biPTH), adjusted serum calcium (Ca), serum phosphorus (P), and calcium-phosphorus product (Ca x P) levels in the management of SHPT in CKD subjects on dialysis by determining achievement of National Kidney Foundation Kidney Disease Outcomes Quality Initiative (K/DOQI) Guideline targets. - To assess the use of vitamin D sterols and phosphate binders when Sensipar is incorporated in the treatment of SHPT. - To assess the safety and tolerability of Sensipar.

ELIGIBILITY:
Inclusion Criteria: - Subjects with chronic kidney disease who have received dialysis for at least one month before the first dose of study medication and are clinically stable. - Adults at least 18 years of age who have given written informed consent. - Out of target PTH values, defined as the most recent historical measurement of biPTH > 160 pg/mL within 3 months prior to informed consent signature. - Serum calcium >/= 8.4 mg/dL within one month prior to informed consent signature. Exclusion Criteria: - Unstable medical condition, defined as having been hospitalized within 30 days before Day 1, or otherwise unstable in the judgement of the investigator. Hospitalization solely for dialysis vascular access revision does not qualify as an unstable medical condition. - Parathyroidectomy in the 3 months before Day 1. - Current gastrointestinal disorder that may be associated with impaired absorption of orally administered medications or an inability to swallow tablets. - Use of investigational drug or device or participation in trial of investigational drug or device (except experimental dialysis machines) within 30 days of enrollment into the study. Any investigational procedures. - Females of child-bearing potential who are pregnant (e.g., positive serum pregnancy test) or are breast feeding. Females of child bearing potential who refuse to use highly effective contraceptive measures (as determined by the investigator) throughout the study. - Hypersensitivity to Sensipar or any of its components. - Previously participated in this or any other Sensipar study, or received/is receiving Sensipar as a commercially available product. - Disorder that would compromise the ability of the subject to give written informed consent and/or to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-07; Study Completion 2005-07

PRIMARY OUTCOMES:
Proportion of subjects with a mean bio-intact parathyroid hormone (biPTH) >/= 80 pg/mL and </= 160 pg/mL (comparable to K/DOQI Guideline target range for intact parathyroid hormone [iPTH] of >/= 150 pg/mL and </= 300 pg/mL) during the assessment phase

SECONDARY OUTCOMES:
Proportion of subjects with mean calcium-phosphorus product (Ca x P) < 55 mgÂ²/dLÂ² during the assessment phase

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_38_AMG_073_20040123.pdf
- See also: FDA-approved Drug Labeling — http://www.sensipar.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com